CLINICAL TRIAL: NCT01549496
Title: A Drug Interaction Study Investigating the Effect of Boceprevir on the Pharmacokinetics of the Calcium Channel Blockers Amlodipine and Diltiazem and Vice Versa in Healthy Volunteers
Brief Title: A Drug Interaction Study of Boceprevir in Combination With Amlodipine or Diltiazem in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator left this hospital
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHRI-BCP-CCB-2012
Record Dates: First submitted 2012-03-01; First posted 2012-03-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Hepatitis C; Hypertension
Keywords: HCV; pharmacokinetics; boceprevir; hypertension; amlodipine; diltiazem
MeSH Terms: conditions — Hepatitis C; Hypertension | interventions — Amlodipine; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- boceprevir (Experimental): boceprevir 800 mg tid
  Interventions: Drug: Amlodipine; Drug: Diltiazem

INTERVENTIONS:
Drug: Amlodipine — amlodipine 2.5 mg QD
Drug: Diltiazem — diltiazem 120 mg qd

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic interactions between the hepatitis C NS3 protease inhibitor boceprevir and the calcium channel blockers amlodipine and diltiazem in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to sign informed consent prior to any study-related activities.
2. Male or female subjects between 18 and 65 years of age inclusive.
3. Healthy, i.e. not suffering from a relevant acute or chronic illness.
4. Body Mass Index (BMI) of 17.5 to 31 kg/m2; and a total body weight > 50 kg (110 lbs).
5. Acceptable medical history, physical examination, and 12-lead ECG at screening.
6. Acceptable laboratory values that indicate adequate baseline organ function at screening visit.
7. Willing to stop using any herbal or natural health products for 2 weeks prior to and during the study including: Grapefruit, grapefruit juice, St. John's Wort.
8. Willingness to abstain from alcohol use for 3 days prior to and during the study.
9. Female subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control:

   * Condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD)
   * A vasectomized partner
   * Total abstinence from sexual intercourse

Exclusion Criteria:

1. Have serological evidence of exposure to HIV or HCV.
2. Known allergies to any of the study medications.
3. Female subjects of childbearing potential who:

   * Has a positive urine pregnancy test at screening.
   * Is not willing to use a reliable method of barrier contraception during the study.
   * Using only oral contraceptive as a birth control method.
   * Is breastfeeding.
4. Inability to adhere to protocol.
5. Use of any medications (2 weeks prior to or during the study) other than occasional use of acetaminophen.
6. Female subjects using contraceptives that contain drospirenone.
7. Subjects that are currently smoking.
8. Subjects with hypertension or heart disease requiring medical treatment.
9. Any condition possibly affecting drug absorption (e.g., gastro intestinal disorder).
10. Patients may be excluded from the study for other reasons, at the investigator's discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
pharmacokinetics | 7 days
  AUC, Cmax, Cmin

SECONDARY OUTCOMES:
number of participants with adverse events | 29 days
  description and frequency of adverse events for all participants during the study

CONTACTS AND LOCATIONS:
Overall Officials: Charles la Porte, PharmD, PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Clinical Investigation Unit, Ottawa Hospital Research Institute, Ottawa, Ontario, Canada